CLINICAL TRIAL: NCT00843505
Title: Telemedicine for Smoking Cessation in Rural Primary Care
Brief Title: Evaluating a Telemedicine Smoking Cessation Program in Rural Primary Care Practices
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kimber Richter, PhD, MPH, MA (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Kimber Richter, PhD, MPH, MA, Associate Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 625; R01HL087643-01A2 (NIH); HL087643-01A2
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Smoking
Keywords: Smoking Cessation; Motivational Interviewing; Quitline; Telemedicine; Stop Smoking Medication
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants will take part in a telemedicine smoking cessation program.
  Interventions: Behavioral: Telemedicine Smoking Cessation Program
- 2 (Active Comparator): Participants will take part in a telephone quitline smoking cessation program.
  Interventions: Behavioral: Telephone Quitline Smoking Cessation Program

INTERVENTIONS:
Behavioral: Telemedicine Smoking Cessation Program — Participants will receive four sessions of telemedicine smoking cessation counseling over an 8-week period. The telemedicine sessions will be delivered by two-way Webcams mounted on desktop computers in the doctors' offices.
  Arms: 1
Behavioral: Telephone Quitline Smoking Cessation Program — Participants will receive four sessions of smoking cessation counseling delivered by telephone in their homes over an 8-week period.
  Arms: 2

SUMMARY:
People who smoke cigarettes and live in rural areas may not have access to a wide variety of resources to help them stop smoking. This study will evaluate two smoking cessation programs-an Internet-based telemedicine program and a telephone-based quitline program-among rural residents.

DETAILED DESCRIPTION:
People who live in rural areas are more likely to smoke cigarettes than people who live in urban and suburban areas. However, many smoking cessation resources and programs may not be available to residents of rural areas. Toll-free tobacco telephone quitlines are proven to help people stop smoking and are available to almost everyone living in the United States, but only 1% to 5% of smokers actually use them. Another option for helping people stop smoking may involve having doctors provide smoking cessation programs in their offices or clinics; however, most doctors' offices do not have the resources to provide this type of service. Telemedicine provides medical information over the phone or through the Internet by using various technologies, including Webcams or video conferencing equipment. It has been used successfully to provide psychiatric care and addictions counseling, but there have been no studies that have examined the effectiveness of a telemedicine smoking cessation program. The purpose of this study is to compare the effectiveness of a telemedicine smoking cessation program that takes place in a doctor's office versus the effectiveness of a traditional telephone quitline smoking cessation program among rural smokers.

The study will be conducted at 25 rural doctors' offices in Kansas. Participants will be randomly assigned to participate in a telephone quitline program or a telemedicine program. Participants in the telephone quitline program will receive four sessions of telephone quitline counseling from smoking cessation counselors over an 8-week period. Participants in the telemedicine program will receive four sessions of telemedicine counseling from smoking cessation counselors over an 8-week period, which will be delivered through two-way Webcams at computers in the doctors' offices. All participants will receive educational handouts and individually tailored quit plans, including information on smoking cessation medications. At baseline and Months 3, 6, and 12, all participants will take part in telephone interviews with study researchers to assess smoking habits. At baseline and Month 12, participants will mail a saliva sample to researchers for the purposes of determining the level of nicotine in the body.

ELIGIBILITY:
Inclusion Criteria:

* Smokes cigarettes every day
* Smokes five or more cigarettes per day
* Has smoked cigarettes for at least 1 year before study entry
* Has a home address and phone number
* Willing to participate in phone assessments
* Willing to be assigned to either of the two study programs

Exclusion Criteria:

* Pregnant or breastfeeding
* Another household member is enrolled in the study
* Moving out of the area of residence in the 14 months after study entry
* Primary care provider is not participating in the study
* Use of other forms of tobacco products (e.g., cigars, spit, snuff) in addition to cigarettes
* Use of a smoking cessation medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 566 (Actual)
Dates: Start 2009-06; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
7-day point prevalence abstinence | Measured at Months 3, 6, and 12

SECONDARY OUTCOMES:
Prolonged abstinence | Measured at Months 3, 6, and 12

CONTACTS AND LOCATIONS:
Overall Officials: Kimber P. Richter, PhD, MPH, MA, Principal Investigator — University of Kansas
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Background] Shireman TI, Tsevat J, Goldie SJ. Time costs associated with cervical cancer screening. Int J Technol Assess Health Care. 2001 Winter;17(1):146-52. doi: 10.1017/s0266462301104137. PMID 11329841
- [Background] Cupertino AP, Mahnken JD, Richter K, Cox LS, Casey G, Resnicow K, Ellerbeck EF. Long-term engagement in smoking cessation counseling among rural smokers. J Health Care Poor Underserved. 2007 Nov;18(4 Suppl):39-51. doi: 10.1353/hpu.2007.0117. PMID 18065851
- [Background] McGinnis JM, Foege WH. Actual causes of death in the United States. JAMA. 1993 Nov 10;270(18):2207-12. PMID 8411605
- [Background] Cronk CE, Sarvela PD. Alcohol, tobacco, and other drug use among rural/small town and urban youth: a secondary analysis of the monitoring the future data set. Am J Public Health. 1997 May;87(5):760-4. doi: 10.2105/ajph.87.5.760. PMID 9184502
- [Background] Doescher MP, Jackson JE, Jerant A, Gary Hart L. Prevalence and trends in smoking: a national rural study. J Rural Health. 2006 Spring;22(2):112-8. doi: 10.1111/j.1748-0361.2006.00018.x. PMID 16606421
- [Background] Stitzer ML. Combined behavioral and pharmacological treatments for smoking cessation. Nicotine Tob Res. 1999;1 Suppl 2:S181-7; discussion S207-10. doi: 10.1080/14622299050012041. PMID 11768178
- [Background] Hughes JR, Goldstein MG, Hurt RD, Shiffman S. Recent advances in the pharmacotherapy of smoking. JAMA. 1999 Jan 6;281(1):72-6. doi: 10.1001/jama.281.1.72. PMID 9892454
- [Background] Silagy C, Lancaster T, Stead L, Mant D, Fowler G. Nicotine replacement therapy for smoking cessation. Cochrane Database Syst Rev. 2004;(3):CD000146. doi: 10.1002/14651858.CD000146.pub2. PMID 15266423
- [Background] Gonzales D, Rennard SI, Nides M, Oncken C, Azoulay S, Billing CB, Watsky EJ, Gong J, Williams KE, Reeves KR; Varenicline Phase 3 Study Group. Varenicline, an alpha4beta2 nicotinic acetylcholine receptor partial agonist, vs sustained-release bupropion and placebo for smoking cessation: a randomized controlled trial. JAMA. 2006 Jul 5;296(1):47-55. doi: 10.1001/jama.296.1.47. PMID 16820546
- [Background] Tonstad S, Tonnesen P, Hajek P, Williams KE, Billing CB, Reeves KR; Varenicline Phase 3 Study Group. Effect of maintenance therapy with varenicline on smoking cessation: a randomized controlled trial. JAMA. 2006 Jul 5;296(1):64-71. doi: 10.1001/jama.296.1.64. PMID 16820548
- [Background] Jorenby DE, Hays JT, Rigotti NA, Azoulay S, Watsky EJ, Williams KE, Billing CB, Gong J, Reeves KR; Varenicline Phase 3 Study Group. Efficacy of varenicline, an alpha4beta2 nicotinic acetylcholine receptor partial agonist, vs placebo or sustained-release bupropion for smoking cessation: a randomized controlled trial. JAMA. 2006 Jul 5;296(1):56-63. doi: 10.1001/jama.296.1.56. PMID 16820547
- [Background] Harris JM Jr. Disease management: new wine in new bottles? Ann Intern Med. 1996 May 1;124(9):838-42. doi: 10.7326/0003-4819-124-9-199605010-00009. PMID 8610954
- [Background] Ockene JK. Physician-delivered interventions for smoking cessation: strategies for increasing effectiveness. Prev Med. 1987 Sep;16(5):723-37. doi: 10.1016/0091-7435(87)90054-5. PMID 3317393
- [Background] Fagerstrom KO. Effects of nicotine chewing gum and follow-up appointments in physician-based smoking cessation. Prev Med. 1984 Sep;13(5):517-27. doi: 10.1016/0091-7435(84)90020-3. PMID 6396639
- [Background] Jamrozik K, Fowler G, Vessey M, Wald N. Placebo controlled trial of nicotine chewing gum in general practice. Br Med J (Clin Res Ed). 1984 Sep 29;289(6448):794-7. doi: 10.1136/bmj.289.6448.794. PMID 6434084
- [Background] Russell MA, Merriman R, Stapleton J, Taylor W. Effect of nicotine chewing gum as an adjunct to general practitioner's advice against smoking. Br Med J (Clin Res Ed). 1983 Dec 10;287(6407):1782-5. doi: 10.1136/bmj.287.6407.1782. PMID 6416593
- [Background] Russell MA, Wilson C, Taylor C, Baker CD. Effect of general practitioners' advice against smoking. Br Med J. 1979 Jul 28;2(6184):231-5. doi: 10.1136/bmj.2.6184.231. PMID 476401
- [Background] Wilson D, Wood G, Johnston N, Sicurella J. Randomized clinical trial of supportive follow-up for cigarette smokers in a family practice. Can Med Assoc J. 1982 Jan 15;126(2):127-9. No abstract available. PMID 7037143
- [Background] Robinson MD, Laurent SL, Little JM Jr. Including smoking status as a new vital sign: it works! J Fam Pract. 1995 Jun;40(6):556-61. PMID 7775909
- [Background] Wechsler H, Levine S, Idelson RK, Rohman M, Taylor JO. The physician's role in health promotion--a survey of primary-care practitioners. N Engl J Med. 1983 Jan 13;308(2):97-100. doi: 10.1056/NEJM198301133080211. No abstract available. PMID 6847940
- [Background] Ockene JK. Smoking intervention: the expanding role of the physician. Am J Public Health. 1987 Jul;77(7):782-3. doi: 10.2105/ajph.77.7.782. No abstract available. PMID 3592029
- [Background] Orleans CT, George LK, Houpt JL, Brodie KH. Health promotion in primary care: a survey of U.S. family practitioners. Prev Med. 1985 Sep;14(5):636-47. doi: 10.1016/0091-7435(85)90083-0. PMID 4070193
- [Background] Wells KB, Lewis CE, Leake B, Schleiter MK, Brook RH. The practices of general and subspecialty internists in counseling about smoking and exercise. Am J Public Health. 1986 Aug;76(8):1009-13. doi: 10.2105/ajph.76.8.1009. PMID 3728756
- [Background] Glasgow RE, Orleans CT, Wagner EH. Does the chronic care model serve also as a template for improving prevention? Milbank Q. 2001;79(4):579-612, iv-v. doi: 10.1111/1468-0009.00222. PMID 11789118
- [Background] Orlandi MA. Promoting health and preventing disease in health care settings: an analysis of barriers. Prev Med. 1987 Jan;16(1):119-30. doi: 10.1016/0091-7435(87)90011-9. PMID 3823010
- [Background] Lewis CE, Wells KB, Ware J. A model for predicting the counseling practices of physicians. J Gen Intern Med. 1986 Jan-Feb;1(1):14-9. doi: 10.1007/BF02596319. PMID 3772565
- [Background] Kottke TE, Battista RN, DeFriese GH, Brekke ML. Attributes of successful smoking cessation interventions in medical practice. A meta-analysis of 39 controlled trials. JAMA. 1988 May 20;259(19):2883-9. doi: 10.1001/jama.259.19.2883. PMID 3367456
- [Background] Epstein RS, Sherwood LM. From outcomes research to disease management: a guide for the perplexed. Ann Intern Med. 1996 May 1;124(9):832-7. doi: 10.7326/0003-4819-124-9-199605010-00008. PMID 8610953
- [Background] Rich MW. Heart failure disease management programs: efficacy and limitations. Am J Med. 2001 Apr 1;110(5):410-2. doi: 10.1016/s0002-9343(01)00632-5. No abstract available. PMID 11286961
- [Background] Rich MW. Heart failure disease management: a critical review. J Card Fail. 1999 Mar;5(1):64-75. doi: 10.1016/s1071-9164(99)90026-x. PMID 10194662
- [Background] Wagner EH. The role of patient care teams in chronic disease management. BMJ. 2000 Feb 26;320(7234):569-72. doi: 10.1136/bmj.320.7234.569. No abstract available. PMID 10688568
- [Background] Wagner EH. Chronic disease management: what will it take to improve care for chronic illness? Eff Clin Pract. 1998 Aug-Sep;1(1):2-4. No abstract available. PMID 10345255
- [Background] Wagner EH, Davis C, Schaefer J, Von Korff M, Austin B. A survey of leading chronic disease management programs: are they consistent with the literature? Manag Care Q. 1999 Summer;7(3):56-66. PMID 10620960
- [Background] Currell R, Urquhart C, Wainwright P, Lewis R. Telemedicine versus face to face patient care: effects on professional practice and health care outcomes. Cochrane Database Syst Rev. 2000;(2):CD002098. doi: 10.1002/14651858.CD002098. PMID 10796678
- [Background] Doolittle GC, Williams AR, Cook DJ. An estimation of costs of a pediatric telemedicine practice in public schools. Med Care. 2003 Jan;41(1):100-9. doi: 10.1097/00005650-200301000-00012. PMID 12544547
- [Background] Stead LF, Perera R, Lancaster T. Telephone counselling for smoking cessation. Cochrane Database Syst Rev. 2006 Jul 19;(3):CD002850. doi: 10.1002/14651858.CD002850.pub2. PMID 16855992
- [Background] Borland R, Segan CJ. The potential of quitlines to increase smoking cessation. Drug Alcohol Rev. 2006 Jan;25(1):73-8. doi: 10.1080/09595230500459537. PMID 16492579
- [Background] Ossip-Klein DJ, McIntosh S. Quitlines in North America: evidence base and applications. Am J Med Sci. 2003 Oct;326(4):201-5. doi: 10.1097/00000441-200310000-00010. PMID 14557735
- [Background] Swartz SH, Cowan TM, Klayman JE, Welton MT, Leonard BA. Use and effectiveness of tobacco telephone counseling and nicotine therapy in Maine. Am J Prev Med. 2005 Nov;29(4):288-94. doi: 10.1016/j.amepre.2005.06.015. PMID 16242591
- [Background] Platt S, Tannahill A, Watson J, Fraser E. Effectiveness of antismoking telephone helpline: follow up survey. BMJ. 1997 May 10;314(7091):1371-5. doi: 10.1136/bmj.314.7091.1371. PMID 9161308
- [Background] Bentz CJ, Bayley KB, Bonin KE, Fleming L, Hollis JF, McAfee T. The feasibility of connecting physician offices to a state-level tobacco quit line. Am J Prev Med. 2006 Jan;30(1):31-7. doi: 10.1016/j.amepre.2005.08.043. PMID 16414421
- [Background] Williams GC, Gagne M, Ryan RM, Deci EL. Facilitating autonomous motivation for smoking cessation. Health Psychol. 2002 Jan;21(1):40-50. PMID 11846344
- [Background] Williams GC, Deci EL. Activating patients for smoking cessation through physician autonomy support. Med Care. 2001 Aug;39(8):813-23. doi: 10.1097/00005650-200108000-00007. PMID 11468500
- [Background] Williams GC, McGregor H, Sharp D, Kouldes RW, Levesque CS, Ryan RM, Deci EL. A self-determination multiple risk intervention trial to improve smokers' health. J Gen Intern Med. 2006 Dec;21(12):1288-94. doi: 10.1111/j.1525-1497.2006.00621.x. PMID 16995893
- [Background] Williams GC, McGregor HA, Sharp D, Levesque C, Kouides RW, Ryan RM, Deci EL. Testing a self-determination theory intervention for motivating tobacco cessation: supporting autonomy and competence in a clinical trial. Health Psychol. 2006 Jan;25(1):91-101. doi: 10.1037/0278-6133.25.1.91. PMID 16448302
- [Background] Burke BL, Arkowitz H, Menchola M. The efficacy of motivational interviewing: a meta-analysis of controlled clinical trials. J Consult Clin Psychol. 2003 Oct;71(5):843-61. doi: 10.1037/0022-006X.71.5.843. PMID 14516234
- [Background] Soria R, Legido A, Escolano C, Lopez Yeste A, Montoya J. A randomised controlled trial of motivational interviewing for smoking cessation. Br J Gen Pract. 2006 Oct;56(531):768-74. PMID 17007707
- [Background] Simon JA, Duncan C, Carmody TP, Hudes ES. Bupropion for smoking cessation: a randomized trial. Arch Intern Med. 2004 Sep 13;164(16):1797-803. doi: 10.1001/archinte.164.16.1797. PMID 15364675
- [Background] Simon JA, Carmody TP, Hudes ES, Snyder E, Murray J. Intensive smoking cessation counseling versus minimal counseling among hospitalized smokers treated with transdermal nicotine replacement: a randomized trial. Am J Med. 2003 May;114(7):555-62. doi: 10.1016/s0002-9343(03)00081-0. PMID 12753879
- [Background] Stephens RS, Roffman RA, Curtin L. Comparison of extended versus brief treatments for marijuana use. J Consult Clin Psychol. 2000 Oct;68(5):898-908. PMID 11068976
- [Background] Stephens RS, Babor TF, Kadden R, Miller M; Marijuana Treatment Project Research Group. The Marijuana Treatment Project: rationale, design and participant characteristics. Addiction. 2002 Dec;97 Suppl 1:109-24. doi: 10.1046/j.1360-0443.97.s01.6.x. PMID 12460133
- [Background] Richter KP, Bammer G. A hierarchy of strategies heroin-using mothers employ to reduce harm to their children. J Subst Abuse Treat. 2000 Dec;19(4):403-13. doi: 10.1016/s0740-5472(00)00137-9. PMID 11166505
- [Background] Richter KP, McCool RM, Okuyemi KS, Mayo MS, Ahluwalia JS. Patients' views on smoking cessation and tobacco harm reduction during drug treatment. Nicotine Tob Res. 2002;4 Suppl 2:S175-82. doi: 10.1080/1462220021000032735. PMID 12573178
- [Background] Richter KP, Kaur H, Resnicow K, Nazir N, Mosier MC, Ahluwalia JS. Cigarette smoking among marijuana users in the United States. Subst Abus. 2004 Jun;25(2):35-43. doi: 10.1300/j465v25n02_06. PMID 15982966
- [Background] Richter KP, Ahluwalia HK, Mosier MC, Nazir N, Ahluwalia JS. A population-based study of cigarette smoking among illicit drug users in the United States. Addiction. 2002 Jul;97(7):861-9. doi: 10.1046/j.1360-0443.2002.00162.x. PMID 12133125
- [Background] Richter KP, McCool RM, Catley D, Hall M, Ahluwalia JS. Dual pharmacotherapy and motivational interviewing for tobacco dependence among drug treatment patients. J Addict Dis. 2005;24(4):79-90. doi: 10.1300/j069v24n04_06. PMID 16368658
- [Background] Jolicoeur DG, Ahluwalia JS, Richter KP, Mosier M, Harris KJ, Gibson C, Moranetz CA. The use of nicotine patches with minimal intervention. Prev Med. 2000 Jun;30(6):504-12. doi: 10.1006/pmed.2000.0670. PMID 10901493
- [Background] Jolicoeur DG, Richter KP, Ahluwalia JS, Mosier MC, Resnicow K. Smoking cessation, smoking reduction, and delayed quitting among smokers given nicotine patches and a self-help pamphlet. Subst Abus. 2003 Jun;24(2):101-6. doi: 10.1080/08897070309511538. PMID 12766377
- [Background] Ahluwalia JS, Richter K, Mayo MS, Ahluwalia HK, Choi WS, Schmelzle KH, Resnicow K. African American smokers interested and eligible for a smoking cessation clinical trial: predictors of not returning for randomization. Ann Epidemiol. 2002 Apr;12(3):206-12. doi: 10.1016/s1047-2797(01)00305-2. PMID 11897179
- [Background] Richter KP, Langel S, Fawcett SB, Paine-Andrews A, Biehler L, Manning R. Promoting the use of advance directives. An empirical study. Arch Fam Med. 1995 Jul;4(7):609-15. doi: 10.1001/archfami.4.7.609. PMID 7606298
- [Background] Richter KP, Surprenant ZJ, Schmelzle KH, Mayo MS. Detecting and documenting intimate partner violence: An intake form question is not enough. Violence Against Women. Vol 9; 2003:458-465.
- [Background] Harris KJ, Richter KP, Schultz J, Johnston J. Formative, process, and intermediate outcome evaluation of a pilot school-based 5 A Day for Better Health Project. Am J Health Promot. 1998 Jul-Aug;12(6):378-81. doi: 10.4278/0890-1171-12.6.378. No abstract available. PMID 10182089
- [Background] Paine-Andrews A, Fawcett SB, Richter KP, Berkley JY, Williams EL, Lopez CM. Community coalition to prevent adolescent substance abuse: The case of the
- [Background] Richter KP, Choi WS, McCool RM, Harris KJ, Ahluwalia JS. Smoking cessation services in U.S. methadone maintenance facilities. Psychiatr Serv. 2004 Nov;55(11):1258-64. doi: 10.1176/appi.ps.55.11.1258. PMID 15534014
- [Background] Ellerbeck EF, Jencks SF, Radford MJ, Kresowik TF, Craig AS, Gold JA, Krumholz HM, Vogel RA. Quality of care for Medicare patients with acute myocardial infarction. A four-state pilot study from the Cooperative Cardiovascular Project. JAMA. 1995 May 17;273(19):1509-14. PMID 7739077
- [Background] Ellerbeck EF, Kresowik TF, Hemann RA, Mason P, Wiblin RT, Marciniak TA. Impact of quality improvement activities on care for acute myocardial infarction. Int J Qual Health Care. 2000 Aug;12(4):305-10. doi: 10.1093/intqhc/12.4.305. PMID 10985268
- [Background] Ellerbeck EF, Totten B, Markello S, Patterson K, Sipe TR, Tilden C. Quality improvement in critical access hospitals: addressing immunizations prior to discharge. J Rural Health. 2003 Fall;19(4):433-8. doi: 10.1111/j.1748-0361.2003.tb00579.x. PMID 14526501
- [Background] Ellerbeck EF. Practice-level variance in ambulatory quality of care. J Gen Intern Med. April 2001 2001;16(supplement 1):192-193.
- [Background] Ellerbeck EF, Choi WS, McCarter K, Jolicoeur DG, Greiner A, Ahluwalia JS. Impact of patient characteristics on physician's smoking cessation strategies. Prev Med. 2003 Apr;36(4):464-70. doi: 10.1016/s0091-7435(02)00055-5. PMID 12649055
- [Background] Engelman KK. Correlates of colorectal cancer screening among Medicare beneficiaries. The Gerontologist. 2000;40 (special issue 1):344
- [Background] Ellerbeck EF, Ahluwalia JS, Jolicoeur DG, Gladden J, Mosier MC. Direct observation of smoking cessation activities in primary care practice. J Fam Pract. 2001 Aug;50(8):688-93. PMID 11509163
- [Background] Engelman KK, Ellerbeck EF, Totten B. Improving systems for preventive care via academic detailing by students. Acad Med. 2001 May;76(5):565-6. doi: 10.1097/00001888-200105000-00115. No abstract available. PMID 11346620
- [Background] Mattioli L, Goertz K, Ardinger R, Belmont J, Cox R, Thomas C. Pediatric cardiology: auscultation from 280 miles away. Kans Med. 1992 Dec;93(12):326, 347-50. PMID 1287282
- [Background] Spaulding RJ, Russo T, Cook DJ, Doolittle GC. Diffusion theory and telemedicine adoption by Kansas health-care providers: critical factors in telemedicine adoption for improved patient access. J Telemed Telecare. 2005;11 Suppl 1:107-9. doi: 10.1258/1357633054461903. PMID 16036015
- [Background] Doolittle GC, Harmon A, Williams A, Allen A, Boysen CD, Wittman C, Mair F, Carlson E. A cost analysis of a tele-oncology practice. J Telemed Telecare. 1997;3 Suppl 1:20-2. doi: 10.1258/1357633971930850. PMID 9218371
- [Background] Cook DJ, Doolittle GC, Ferguson D, Hanks N, Hood J, Howard M, Troha J, Mehling D, Zurbuchen N. Explaining the adoption of telemedicine services: an analysis of a paediatric telemedicine service. J Telemed Telecare. 2002;8 Suppl 2:106-7. doi: 10.1177/1357633X020080S248. PMID 12217159
- [Background] Doolittle GC, Williams AR, Spaulding A, Spaulding RJ, Cook DJ. A cost analysis of a tele-oncology practice in the United States. J Telemed Telecare. 2004;10 Suppl 1:27-9. doi: 10.1258/1357633042614429. PMID 15603601
- [Background] Zink T, Shireman T. Teen compliance with contraception. Analysis Of the ohio medicaid claims data. J Pediatr Adolesc Gynecol. 2000 May;13(2):97. doi: 10.1016/s1083-3188(00)00035-8. PMID 10869992
- [Background] Shireman TI, Heaton PC, Gay WE, Cluxton RJ, Moomaw CJ. Relationship between asthma drug therapy patterns and healthcare utilization. Ann Pharmacother. 2002 Apr;36(4):557-64. doi: 10.1345/aph.1A067. PMID 11918499
- [Background] Zink TM, Shireman TI, Ho M, Buchanan T. High-risk teen compliance with prescription contraception: an analysis of Ohio Medicaid claims. J Pediatr Adolesc Gynecol. 2002 Feb;15(1):15-21. doi: 10.1016/s1083-3188(01)00134-6. PMID 11888805
- [Background] Svarstad BL, Shireman TI, Sweeney JK. Using drug claims data to assess the relationship of medication adherence with hospitalization and costs. Psychiatr Serv. 2001 Jun;52(6):805-11. doi: 10.1176/appi.ps.52.6.805. PMID 11376229
- [Background] Shireman TI, Hall JP, Rigler SK, Moore JM. Medicaid's expenditures for newer pharmacotherapies for adults with disabilities. Health Care Financ Rev. 2007 Summer;28(4):31-41. PMID 17722749
- [Background] Richter KP, Hamilton AK, Hall S, Catley D, Cox LS, Grobe J. Patterns of smoking and methadone dose in drug treatment patients. Exp Clin Psychopharmacol. 2007 Apr;15(2):144-53. doi: 10.1037/1064-1297.15.2.144. PMID 17469938
- [Background] Harris KJ, Ahluwalia JS, Catley D, Okuyemi KS, Mayo MS, Resnicow K. Successful recruitment of minorities into clinical trials: The Kick It at Swope project. Nicotine Tob Res. 2003 Aug;5(4):575-84. doi: 10.1080/1462220031000118540. PMID 12959796
- [Background] Ahluwalia JS, Harris KJ, Catley D, Okuyemi KS, Mayo MS. Sustained-release bupropion for smoking cessation in African Americans: a randomized controlled trial. JAMA. 2002 Jul 24-31;288(4):468-74. doi: 10.1001/jama.288.4.468. PMID 12132977
- [Background] Catley D, Harris KJ, Okuyemi KS, Mayo MS, Pankey E, Ahluwalia JS. The influence of depressive symptoms on smoking cessation among African Americans in a randomized trial of bupropion. Nicotine Tob Res. 2005 Dec;7(6):859-70. doi: 10.1080/14622200500330118. PMID 16298721
- [Background] Boardman T, Catley D, Mayo MS, Ahluwalia JS. Self-efficacy and motivation to quit during participation in a smoking cessation program. Int J Behav Med. 2005;12(4):266-72. doi: 10.1207/s15327558ijbm1204_7. PMID 16262545
- [Background] Manning BK, Catley D, Harris KJ, Mayo MS, Ahluwalia JS. Stress and quitting among African American smokers. J Behav Med. 2005 Aug;28(4):325-33. doi: 10.1007/s10865-005-9004-9. PMID 16049631
- [Background] Nollen NL, Catley D, Davies G, Hall M, Ahluwalia JS. Religiosity, social support, and smoking cessation among urban African American smokers. Addict Behav. 2005 Jul;30(6):1225-9. doi: 10.1016/j.addbeh.2004.10.004. Epub 2004 Nov 10. PMID 15925130
- [Background] Lee RE, Harris KJ, Catley D, Shostrom V, Choi S, Mayo MS, Okuyemi K, Kaur H, Ahluwalia JS. Factors associated with BMI, weight perceptions and trying to lose weight in African-American smokers. J Natl Med Assoc. 2005 Jan;97(1):53-61. PMID 15719872
- [Background] Pulvers KM, Catley D, Okuyemi K, Scheibmeir M, McCarter K, Jeffries SK, Ahluwalia JS. Gender, smoking expectancies, and readiness to quit among urban African American smokers. Addict Behav. 2004 Aug;29(6):1259-63. doi: 10.1016/j.addbeh.2004.03.028. PMID 15236832
- [Background] Boardman T, Catley D, Grobe JE, Little TD, Ahluwalia JS. Using motivational interviewing with smokers: do therapist behaviors relate to engagement and therapeutic alliance? J Subst Abuse Treat. 2006 Dec;31(4):329-39. doi: 10.1016/j.jsat.2006.05.006. Epub 2006 Aug 1. PMID 17084786
- [Background] Cupertino PA, Richter KP, Cox LS, Nazir N, Greiner AK, Ahluwalia JS, Ellerbeck EF. Smoking cessation pharmacotherapy preferences in rural primary care. Nicotine Tob Res. 2008 Feb;10(2):301-7. doi: 10.1080/14622200701825817. PMID 18236294
- [Background] Greiner KA, Engelman KK, Hall MA, Ellerbeck EF. Barriers to colorectal cancer screening in rural primary care. Prev Med. 2004 Mar;38(3):269-75. doi: 10.1016/j.ypmed.2003.11.001. PMID 14766108
- [Background] Engelman KK, Perpich DL, Peterson SL, Hall MA, Ellerbeck EF, Stanton AL. Cancer information needs in rural areas. J Health Commun. 2005 Apr-May;10(3):199-208. doi: 10.1080/10810730590934217. PMID 16036728
- [Background] Anis NA, Lee RE, Ellerbeck EF, Nazir N, Greiner KA, Ahluwalia JS. Direct observation of physician counseling on dietary habits and exercise: patient, physician, and office correlates. Prev Med. 2004 Feb;38(2):198-202. doi: 10.1016/j.ypmed.2003.09.046. PMID 14715212
- [Background] Miller WR, Benefield RG, Tonigan JS. Enhancing motivation for change in problem drinking: a controlled comparison of two therapist styles. J Consult Clin Psychol. 1993 Jun;61(3):455-61. doi: 10.1037//0022-006x.61.3.455. PMID 8326047
- [Background] Etter JF, Neidhart E, Bertrand S, Malafosse A, Bertrand D. Collecting saliva by mail for genetic and cotinine analyses in participants recruited through the Internet. Eur J Epidemiol. 2005;20(10):833-8. doi: 10.1007/s10654-005-2148-7. PMID 16283473
- [Background] Hughes JR, Keely JP, Niaura RS, Ossip-Klein DJ, Richmond RL, Swan GE. Measures of abstinence in clinical trials: issues and recommendations. Nicotine Tob Res. 2003 Feb;5(1):13-25. PMID 12745503
- [Background] SRNT Subcommittee on Biochemical Verification. Biochemical verification of tobacco use and cessation. Nicotine Tob Res. 2002 May;4(2):149-59. doi: 10.1080/14622200210123581. No abstract available. PMID 12028847
- [Background] Spierto FW, Hannon WH, Kendrick JS, Bernert JT, Pirkle JL, Gargiullo P. Urinary cotinine levels in women enrolled in a smoking cessation study during and after pregnancy. J Smoking-Related Dis. 1988;5(2):65-76.
- [Background] Jacob P 3rd, Wilson M, Benowitz NL. Improved gas chromatographic method for the determination of nicotine and cotinine in biologic fluids. J Chromatogr. 1981 Jan 2;222(1):61-70. doi: 10.1016/s0378-4347(00)81033-6. PMID 6783675
- [Background] Hyland A, Cummings KM, Lynn WR, Corle D, Giffen CA. Effect of proxy-reported smoking status on population estimates of smoking prevalence. Am J Epidemiol. 1997 Apr 15;145(8):746-51. doi: 10.1093/aje/145.8.746. PMID 9126001
- [Background] Gilpin EA, Pierce JP, Cavin SW, Berry CC, Evans NJ, Johnson M, Bal DG. Estimates of population smoking prevalence: self-vs proxy reports of smoking status. Am J Public Health. 1994 Oct;84(10):1576-9. doi: 10.2105/ajph.84.10.1576. PMID 7943473
- [Background] Chen Y, Rennie DC, Dosman JA. The reliability of cigarette consumption reports by spousal proxies. Am J Public Health. 1995 Dec;85(12):1711-2. doi: 10.2105/ajph.85.12.1711. No abstract available. PMID 7503354
- [Background] Ryan RM, Connell JP. Perceived locus of causality and internalization: examining reasons for acting in two domains. J Pers Soc Psychol. 1989 Nov;57(5):749-61. doi: 10.1037//0022-3514.57.5.749. PMID 2810024
- [Background] Pbert L, Adams A, Quirk M, Hebert JR, Ockene JK, Luippold RS. The patient exit interview as an assessment of physician-delivered smoking intervention: a validation study. Health Psychol. 1999 Mar;18(2):183-8. doi: 10.1037//0278-6133.18.2.183. PMID 10194054
- [Background] Royce JM, Hymowitz N, Corbett K, Hartwell TD, Orlandi MA. Smoking cessation factors among African Americans and whites. COMMIT Research Group. Am J Public Health. 1993 Feb;83(2):220-6. doi: 10.2105/ajph.83.2.220. PMID 8427327
- [Background] Fagerstrom KO, Schneider NG. Measuring nicotine dependence: a review of the Fagerstrom Tolerance Questionnaire. J Behav Med. 1989 Apr;12(2):159-82. doi: 10.1007/BF00846549. PMID 2668531
- [Background] Katon W, Schulberg H. Epidemiology of depression in primary care. Gen Hosp Psychiatry. 1992 Jul;14(4):237-47. doi: 10.1016/0163-8343(92)90094-q. PMID 1505745
- [Background] Irwin M, Artin KH, Oxman MN. Screening for depression in the older adult: criterion validity of the 10-item Center for Epidemiological Studies Depression Scale (CES-D). Arch Intern Med. 1999 Aug 9-23;159(15):1701-4. doi: 10.1001/archinte.159.15.1701. PMID 10448771
- [Background] Glassman AH. Cigarette smoking: implications for psychiatric illness. Am J Psychiatry. 1993 Apr;150(4):546-53. doi: 10.1176/ajp.150.4.546. PMID 8465868
- [Background] Barry KL, Fleming MF. The Alcohol Use Disorders Identification Test (AUDIT) and the SMAST-13: predictive validity in a rural primary care sample. Alcohol Alcohol. 1993 Jan;28(1):33-42. PMID 8471085
- [Background] Isaacson JH, Butler R, Zacharek M, Tzelepis A. Screening with the Alcohol use Disorders Identification Test (AUDIT) in an inner-city population. J Gen Intern Med. 1994 Oct;9(10):550-3. doi: 10.1007/BF02599279. PMID 7823225
- [Background] Hays RD, Sherbourne CD, Mazel RM. The RAND 36-Item Health Survey 1.0. Health Econ. 1993 Oct;2(3):217-27. doi: 10.1002/hec.4730020305. PMID 8275167
- [Background] Ludwig DS. The glycemic index: physiological mechanisms relating to obesity, diabetes, and cardiovascular disease. JAMA. 2002 May 8;287(18):2414-23. doi: 10.1001/jama.287.18.2414. PMID 11988062
- [Background] Hoyle RH, Kenny DA. Sample size, reliability, and tests of statistical mediation. In: Hoyle RH, ed. Statistical strategies for small sample research. Thousand Oaks, CA: Sage; 1999
- [Background] Stone CA, Sobel ME. The robustness of estimates of total indirect effects in covariance structure models estimated by maximum likelihood. Psychometrika. 1990;55(337-52).
- [Background] Kenny DA, Kashy DA, Bolger N. Data analysis in social psychology. In: Gilbert DT, Fiske ST, Lindzey G, eds. The Handbook of Social Psychology, Volume 1. New York: Oxford University Press; 1998:233-265
- [Background] Preacher KJ, Hayes AF. SPSS and SAS procedures for estimating indirect effects in simple mediation models. Behav Res Methods Instrum Comput. 2004 Nov;36(4):717-31. doi: 10.3758/bf03206553. PMID 15641418
- [Background] MacKinnon DP, Lockwood CM, Hoffman JM, West SG, Sheets V. A comparison of methods to test mediation and other intervening variable effects. Psychol Methods. 2002 Mar;7(1):83-104. doi: 10.1037/1082-989x.7.1.83. PMID 11928892
- [Background] Curry SJ, McBride C, Grothaus LC, Louie D, Wagner EH. A randomized trial of self-help materials, personalized feedback, and telephone counseling with nonvolunteer smokers. J Consult Clin Psychol. 1995 Dec;63(6):1005-14. doi: 10.1037//0022-006x.63.6.1005. PMID 8543703
- [Background] Aveyard P, Griffin C, Lawrence T, Cheng KK. A controlled trial of an expert system and self-help manual intervention based on the stages of change versus standard self-help materials in smoking cessation. Addiction. 2003 Mar;98(3):345-54. doi: 10.1046/j.1360-0443.2003.00302.x. PMID 12603234
- [Background] Glaser B, Strauss A. The Discovery of Grounded Theory: Strategies for Qualitative Research. Chicago: Aldine; 1967
- [Background] Winer BJ. Statistical principles in experiemntal design. (2nd Edition): New York: McGraw-Hill; 1971
- [Background] Baron RM, Kenny DA. The moderator-mediator variable distinction in social psychological research: conceptual, strategic, and statistical considerations. J Pers Soc Psychol. 1986 Dec;51(6):1173-82. doi: 10.1037//0022-3514.51.6.1173. PMID 3806354
- [Background] Brown RL. Assessing specific mediational effects in complex theoretical models. Structural Equation Modeling. 1997;4:142-156
- [Background] Shrout PE, Bolger N. Mediation in experimental and nonexperimental studies: new procedures and recommendations. Psychol Methods. 2002 Dec;7(4):422-45. PMID 12530702
- [Background] Gold MR. Cost-effectiveness in health and medicine. New York: Oxford University Press; 1996.
- [Background] Haddix AC, Teutsch SM, Corso PS. Prevention effectiveness: a guide to decision analysis and economic evaluation. 2nd ed. Oxford ; New York: Oxford University Press; 2003.
- [Background] Parrott S, Godfrey C, Raw M, West R, McNeill A. Guidance for commissioners on the cost effectiveness of smoking cessation interventions. Thorax. 1998 Dec;53 Suppl 5 Pt 2(Suppl 5):S1-38. No abstract available. PMID 10226676
- [Background] Tengs TO, Adams ME, Pliskin JS, Safran DG, Siegel JE, Weinstein MC, Graham JD. Five-hundred life-saving interventions and their cost-effectiveness. Risk Anal. 1995 Jun;15(3):369-90. doi: 10.1111/j.1539-6924.1995.tb00330.x. PMID 7604170
- [Background] Miller WR, Rollnick S. Motivational interviewing: Preparing people to change addictive behavior. New York: Guilford Press; 1991.
- [Background] Centers for Disease Control and Prevention (CDC). State-specific prevalence of current cigarette smoking among adults and secondhand smoke rules and policies in homes and workplaces--United States, 2005. MMWR Morb Mortal Wkly Rep. 2006 Oct 27;55(42):1148-51. PMID 17065980
- [Background] American Medical Association. Physician Characteristics and Distribution in the US, 2007. Chicago, IL: American Medical Association; 2007.
- [Background] Cupertino AP, Richter KP, Ellerbeck EF, Cox LS, Spaulding R. A Pilot study of telemedicine for smoking cessation Society for Research on Nicotine and Tobacco. Orlando - FL; 2006.
- [Background] Doolittle GL, Spaulding A, Spaulding RJ. The financial side of a tele-oncology practice. In: Whitten P, Cook DJ, eds. Understanding Health Communication Technologies. San Francisco - CA: Jossey-Bass; 2004.
- [Background] Nelson EL, Spaulding RJ. Adapting a patient-provider interaction coding system for interactive televideo. 2004;10:73.
- [Background] Miller WR, Rollnick S. Motivational Interviewing: Preparing people for change. 2nd ed. ed. New York: Guilford Press; 2002.
- [Background] Miller W. Combined Behavioral Intervention Manual: A Clinical Research Guide for Therapists Treating People with Alcohol Abuse and Dependence. DHHS Publication No. (NIH) 04-5288. Vol Volume 1. Bethesda, MD: DHHS Publication No. (NIH) 04-5288; 2004.
- [Background] Bedrosian RC, Beck AT. Principles of cognitive therapy. In: Mahoney MH, ed. Psychotherapy Process: Current Issues and Future Directions. New York: Plenum; 1980:127-152.
- [Background] Beck AT. Cognitive Therapy. In: Kaplan HI, Sadock BJ, eds. Comprehensive Textbook of Psychiatry. Vol II. New York: Williams and Wilkins; 1985:1432-1438.
- [Background] Markland D, Ryan RM, Tobin VJ, Rollnick S. Motivational Interviewing and Self-Determination Theory. Journal of Social and Clinical Psychology. 2005;24(6):811-831.
- [Background] Deci EL, Ryan RM. Handbook of self-determination research. Rochester, NY: University of Rochester Press; 2002.
- [Background] Deci EL, Ryan RM. Intrinsic motivation and self-determination in human behavior. New York: Plenum; 1985.
- [Background] Centers for Medicare & Medicaid Services. Medicare Benefit Policy Manual: Chapter 15 - Covered Medical and Other Health Services. Revision 37 ed: Centers for Medicare & Medicaid Services; 2005.
- [Background] Centers for Disease Control and Prevention (CDC). Physician and other health-care professional counseling of smokers to quit--United States, 1991. MMWR Morb Mortal Wkly Rep. 1993 Nov 12;42(44):854-7. PMID 8232167
- [Background] Fiore MC, Bailey WC, Cohen SJ, al. et. Treating Tobacco Use and Dependence. Clinical Practice Guideline. Rockville, MD: U.S. Department of Health and Human Services. Public Health Service.; 2000.
- [Background] Kansas Department of Health and Environment. Primary Care: Health Professional Underserved Areas Report. Office of Local and Rural Health; 2004.
- [Background] Eberhardt MS, Ingram DD, Makuc D. Urban and Rural Health Chartbook: Health United States, 2001. Hyattsville, MD: National Center for Health Statistics; 2001.
- [Background] Centers for Disease Control (CDC). Cigarette smoking among adults--United States, 1988. MMWR Morb Mortal Wkly Rep. 1991 Nov 8;40(44):757-9, 765. PMID 1944122
- [Background] Centers for Disease Control and Prevention (CDC). Tobacco use among adults--United States, 2005. MMWR Morb Mortal Wkly Rep. 2006 Oct 27;55(42):1145-8. PMID 17065979
- [Background] Bailey L. An Overview of NAQC. National Network of Tobacco Cessation Quitlines 2006 Regional Meeting -- Western Region. San Diego, CA; 2006.
- [Background] Levin HM, McEwan PJ. Cost-effectiveness analysis: Methods and applications. 2nd ed. Thousand Oaks, Calif.: Sage Publications; 2001.
- [Background] Moyers TB, Martin T, Manuel JK, Miller WR, Ernst D. Revised Global Scales: Motivational Interviewing Treatment Integrity (MITI) 3.0: University of New Mexico Center on Alcoholism, Substance Abuse and Addictions (CASAA); 2007.
- [Background] Staines GL. Comparative outcome evaluations of psychotherapies: Guidelines for addressing eight limitations of the gold standard of causal inference. Psychotherapy (Chic). 2007 Jun;44(2):161-74. doi: 10.1037/0033-3204.44.2.161. PMID 22122208
- [Derived] Richter KP, Shireman TI, Ellerbeck EF, Cupertino AP, Catley D, Cox LS, Preacher KJ, Spaulding R, Mussulman LM, Nazir N, Hunt JJ, Lambart L. Comparative and cost effectiveness of telemedicine versus telephone counseling for smoking cessation. J Med Internet Res. 2015 May 8;17(5):e113. doi: 10.2196/jmir.3975. PMID 25956257
- [Derived] Mussulman L, Ellerbeck EF, Cupertino AP, Preacher KJ, Spaulding R, Catley D, Cox LS, Lambart L, Hunt JJ, Nazir N, Shireman T, Richter KP. Design and participant characteristics of a randomized-controlled trial of telemedicine for smoking cessation among rural smokers. Contemp Clin Trials. 2014 Jul;38(2):173-81. doi: 10.1016/j.cct.2014.04.008. Epub 2014 Apr 24. PMID 24768940
- See also: Click here for the "Telemedicine: Past, Present, Future" article Web page. — http://www.nlm.nih.gov/archive/20040830/pubs/cbm/telembib.html
- See also: Click here for the Telecommunications Service in Rural America Web page on the Federal Communications Commission Web site. — http://www.fcc.gov/cgb/rural
- See also: Click here for the North American Quitline Consortium, part of the National Cancer Institute, "1-800-Quit Now" Data for U.S. States (Available to members or by e-mail request to: NAQC@americanlegacy.org) — http://www.naquitline.org/
- See also: Click here for the Center for Tobacco Research and Intervention Fact Sheets Web site. — http://www.ctri.wisc.edu/News.Center/News.Center_FactSheets.html